CLINICAL TRIAL: NCT04690673
Title: Detection of Paracetamol Concentration in Blood-, Saline- and Urine Samples With an Electrochemical Indicator in Healthy Volunteers - a Validation Study for a Novel Technique
Brief Title: Detection of Paracetamol Concentration in Blood-, Saline- and Urine Samples - a Validation Study for a Novel Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johanna Kujala (Other)
Responsible Party: Sponsor-Investigator, Johanna Kujala, Sponsor-Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FEPODPara2020-1
Record Dates: First submitted 2020-12-14; First posted 2020-12-31 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Drug Mechanism; Healthy
Keywords: electrochemical; Paracetamol; Lipidomics; Endocannabinoid system
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): All healthy volunteers are in this group. They receive 1g paracetamol orally. Saline-, urine-, venous blood and fingerprick samples will be collected at timely intervals.
  Interventions: Drug: Paracetamol; Diagnostic Test: Paracetamol concentration measurements and lipidomic assessment

INTERVENTIONS:
Drug: Paracetamol — 1 g oral paractamol
Diagnostic Test: Paracetamol concentration measurements and lipidomic assessment — Paracetamol concentration is measured from saline-, urine-, venous blood- and fingerprick- samples at timely intervals. Also serum lipidomic assessment is performed from venous blood samples.

SUMMARY:
The main objective is to assess whether a novel electrochemical tool is reliable in detecting concentration of paracetamol in fingerprick- , saline-, urine-, and serum samples. We will recruit 12 healthy volunteers aged 18-45. They will get 1 g oral paracetamol. Paracetamol concentration will be detected from abovementioned samples at timely intervals for 24 hours, analyzed with the novel electrochemical method and compared to gold standard mass-spectrometry analysis.

Despite of extensive use, the mechanism of action of parasetamol is not completely understood. The central serotonergic system may play a role. Endocannabinoid system is a group of lipid mediators, that possibly is involved in mediating paracetamol effect to the serotonergic system. Serum lipidomic assessment can be used to study endocannabinoid metabolics. In this study we will try to assess changes in endocannabinoid system by looking into serum lipidomics in order to understand the mechanism of action of paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, no medication of any kind.
* Age 18-45
* BMI 18.5 - 30
* Informed consent

Exclusion Criteria:

* Pregnancy, lactation.
* prisoner
* smoking
* less than 3 months from prior blood donation or clinical pharmacological study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki university hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was announced on Helsinki University student's website in January 2021.
Pre-assignment Details: No medications or nutritional supplements were allowed prior to the study day.
Period: Overall Study
Arm/Group | Study Group
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Finland | 12

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Geometric Means of Cmax and AUC 0-last of Paracetamol Measured by the Novel Electrochemical Method With Mass-spectrometry in Capillary Whole Blood Samples.
Description: Geometric mean values of the highest paracetamol concentrations (Cmax) and area under the curve (AUC) measured with the novel electrochemical method were compared with the 'gold standard' mass-spectrometry (control) from capillary whole blood samples. The data are presented as the ratio of geometric means to control, geometric coefficients of variation (as percentage) as a measure of dispersion.
Time Frame: 1 day
Population: All healthy volunteers in this group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio-to-control
Groups:
- Cmax: Comparison of the geometric mean values of the maximum capillary paracetamol concentrations (Cmax) measured with the electrochemical method and the mass-spectrometry (control). Data are presented as ratio-to-control.
- AUC 0-last: Comparison of the geometric means of the area- under-the-curve (AUC) from timepoints 0-last measured with the electrochemical method and the mass-spectrometry (control). Data are presented as ratio-to-control.
Arm/Group | Cmax | AUC 0-last
Number analyzed (Participants) | 12 | 12
ratio-to-control | 1.03 (21) | 1.17 (29)
Statistical Analysis 1: Comparison: Cmax; Highest paracetamol concentrations (Cmax) measured from capillary with the electrochemical method compared with measurements with mass-spectrometry; Test type: Equivalence — Based on previous reports on the pharmacokinetics of oral paracetamol, the standard deviation of the within-subject difference in the Cmax for paracetamol was estimated to be 35% of the mean Cmax. Using this standard deviation, 10 participants were estimated to be sufficient, with a power of at least 80% (at 5% significance level). We recruited 12 volunteers to account for potential protocol violations or dropouts; p = 0.05, t-test, 2 sided — Not adjusted for multiple comparisons as the analysis was exploratory; Geometric mean ratio = 1.03, 90% CI 2-sided [0.94 to 1.13] — Adhering

2. Secondary Outcome: Comparison of Geometric Means of Cmax and AUC 0-last of Paracetamol in Capillary With Venous Plasma (Control), Both Measured by Mass-spectrometry.
Description: Geometric mean values of the highest paracetamol concentrations (Cmax) and area under the curve -calculations (AUC0-last) measured by mass-spectrometry were compared between capillary and plasma (control) to analyse paracetamol pharmacokinetics. The data are presented as ratio-to-control with geometric coefficients of variation (as percentage).
Time Frame: 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio-to-control
Groups:
- Cmax: Comparison of the geometric means of the highest paracetamol concentrations (Cmax) measured in capillary and venous plasma (control), both measurements were performed by mass-spectrometry. The data are presented as ratio-to-control with geometric coefficients of variation (as percentage).
- AUC 0-last: Comparison of the geometric means of the area- under-the-curve (AUC) from timepoints 0-last measured from capillary and venous plasma (control). Data are presented as ratio-to-control with geometric coefficients of variation (as percentage).
Arm/Group | Cmax | AUC 0-last
Number analyzed (Participants) | 12 | 12
ratio-to-control | 1.50 (31) | 1.08 (30)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT04690673/Prot_SAP_000.pdf